CLINICAL TRIAL: NCT05322785
Title: Optimization of Exhaled Biomarker Collection and Analysis
Acronym: EBC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Michael D. Davis, Assistant Research Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1910580775
Record Dates: First submitted 2022-03-14; First posted 2022-04-12 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Disease; Healthy
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Intervention Model Description: Study sample will consist of individuals aged 4-110 with a diagnosis of acute or chronic respiratory disorders, or metabolic or systemic conditions involving diffuse inflammation, or normal subjects with no pulmonary disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Visit breath collection (Other): Following informed consent, exhaled breath will be passively collected from subjects during quiet oral breathing through a simple mouthpiece or mask. Exhaled breath will be diverted into a collection device, which may include a bag, tube, or other device with minimal resistance. The collection process, including completing forms, will not exceed 30 minutes.
  At no time will the patients be breathing anything other than ambient air with or without oxygen enrichment as clinically indicated. Inhaled air will not be manipulated.
  Interventions: Other: Breath collection

INTERVENTIONS:
Other: Breath collection — Exhaled breath will be passively collected from subjects during quiet oral breathing through a simple mouthpiece or mask

SUMMARY:
This is an exploratory study designed to optimize, standardize, and validate novel breath biomarkers; there are no objective endpoints. The goal of this study is to generate pilot data to be used to generate hypothesis-driven studies.

DETAILED DESCRIPTION:
Exhaled breath has three fractions - gaseous breath, volatile breath, and breath condensate. Biomarkers have been identified in each of these fractions and non-invasive collection methods have been developed. Exhaled breath can be safely and easily performed in all patient populations, including neonatal children and the elderly. We have shown that relative to normal controls, condensed exhalates obtained from asthmatic subjects reproducibly contain elevated concentrations of oxides of nitrogen and are more acidic (having hydrogen ion concentrations two to three log orders higher). We wish to extend these studies across all breath fractions and other lung diseases and respiratory processes including viral upper respiratory tract infections, cystic fibrosis, pneumonia, pulmonary hypertension, bronchiolitis obliterans, chronic obstructive pulmonary disease, tracheostomized patients and cigarette smokers. Through this study extension, we will obtain pilot data/preliminary information about the potential utility of this new technique to non-invasively evaluate disease status in various respiratory diseases. We also wish to obtain data regarding specificity by evaluating the exhaled breath obtained from patients with non-respiratory illnesses, such as, but not limited to diabetes, gastroenteritis, and various inflammatory disorders. We think it is likely that the exhaled biomarkers reflect underlying airway inflammation and infection.

Following informed consent, exhaled breath will be passively collected from subjects during quiet oral breathing through a simple mouthpiece or mask. Exhaled breath will be diverted into a collection device, which may include a bag, tube, or other device with minimal resistance. The collection process, including completing forms, will not exceed 30 minutes.

Subjects may be asked to provide several specimens during the course of their inpatient stay or clinic visit to obtain longitudinal data.

At no time will the patients be breathing anything other than ambient air with or without oxygen enrichment as clinically indicated. Inhaled air will not be manipulated.

Exhaled breath collection technique is completely comfortable, causing neither discomfort nor fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Study sample will consist of individuals aged 4-110 with a diagnosis of acute or chronic respiratory disorders, or metabolic or systemic conditions involving diffuse inflammation, or normal subjects with no pulmonary disease.

Exclusion Criteria:

* Subjects that are unable or unwilling to cooperate with specimen collection.

Ages: 4 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-02-02 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Breath amount, pH, components | During the exhaled breath collection procedure, not to exceed 30 minutes
  Breath collected will be measured for total volume of condensation collected, pH from the pH scale and other components of airway factors

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine - Wells Center for Pediatric Research, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis MD, Fowler SJ, Montpetit AJ. Exhaled breath testing - A tool for the clinician and researcher. Paediatr Respir Rev. 2019 Feb;29:37-41. doi: 10.1016/j.prrv.2018.05.002. Epub 2018 May 17. PMID 29921519
- [Background] Davis MD, Montpetit AJ. Exhaled Breath Condensate: An Update. Immunol Allergy Clin North Am. 2018 Nov;38(4):667-678. doi: 10.1016/j.iac.2018.06.002. Epub 2018 Sep 21. PMID 30342587
- [Background] Vaughan J, Ngamtrakulpanit L, Pajewski TN, Turner R, Nguyen TA, Smith A, Urban P, Hom S, Gaston B, Hunt J. Exhaled breath condensate pH is a robust and reproducible assay of airway acidity. Eur Respir J. 2003 Dec;22(6):889-94. doi: 10.1183/09031936.03.00038803. PMID 14680074